CLINICAL TRIAL: NCT02983136
Title: Safe Hands at the Sharp End- Implementing Aseptic Technique in the Operating Room, A Prospective Controlled Study With an Embedded Process Evaluation
Brief Title: Safe Hands at the Sharp End- Implementing Aseptic Technique in the Operating Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: University of Gothenburg Center for Person-Centred Care, GPCC (Unknown); Landstingens Ömsesidiga Försäkringsbolag (Löf) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Safe Hands
Record Dates: First submitted 2016-11-28; First posted 2016-12-06 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Surgical Wound Infection
Keywords: Hand Hygiene; Implementation; Partnership; Surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study site (Experimental): The study arm will consist of managers and staff at at the operating department of a University hospital in western Sweden' The intervention is based on partnership, dialogue and inter-professional learning
  Interventions: Behavioral: Dialogue and inter-professional learning
- Control site (No Intervention): The Control arm will consist of managers and staff at at the operating department of a University hospital in south Sweden

INTERVENTIONS:
Behavioral: Dialogue and inter-professional learning — The middle and front-line leaders of the study OR will participate in an intervention based on an iKT model. Components of the intervention will include:
  * Two workshops, consisting of educational sessions covering the state of the art regarding person-centeredness, prevention of infections, leadership, and implementation. The educational component and results of pre-studies will work as frameworks for the dialogues between the front-line leaders and the research group. In dialogues the participants will be given the opportunity to reflect on barriers to and enablers of change; and
  * The participants will be supported in creating an action plan aimed at facilitating the anaesthesia providers' change of practice.
  Arms: Study site

SUMMARY:
The aim of this integrated Knowledge Translation (iKT) study is to develop and test a multifaceted implementation intervention for feasibility, acceptability and effectiveness. The intervention will be tailored to fit the context of the operating room (OR), to promote OR team members' use of aseptic techniques during the care of frail persons undergoing acute fracture surgery of the hip.

Through the use of an iKT approach, the investigators hypothesise that building on leadership support, partnership between researchers, managers/clinical leaders and healthcare professionals, a solid foundation for the sustained implementation of patient safety innovations can be created.

DETAILED DESCRIPTION:
PROJECT DESCRIPTION

Aim The aim of this iKT study is to develop and test a multifaceted implementation intervention for feasibility, acceptability and effectiveness.The intervention will be tailored to fit the inner context of the operating department, to promote anaesthetic providers use of aseptic techniques.

Theory In designing the present study, the investigators followed the four iterative phases as identified by the UK Medical Research Council (MRC) framework for developing and evaluating complex interventions(1): *Review of the theoretical basis for the innovation and the context *Conducting pre studies and designing the intervention,*The exploratory trial i.e. the intervention implementation and evaluation.

The aim of the leadership intervention is to support the leaders in developing a participatory and effective leadership behaviours that promote the OR team's use of aseptic techniques and facilitate inter professional learning. The middle and front-line leaders of the study OR will participate in an intervention based on an iKT model inspired by person-centeredness (2) social construction and complexity thinking (3). The care professionals participating in this in this study are considered active partners and co-creators of the implementation process and activities. This type of collaborative approach means that the researchers, leaders and the OR team work closely together throughout the research process in order to produce findings that are relevant for users and context (4). Using this innovative approach represents a major departure from the concept of 'compliance' and a shift towards change as a result of a participatory and mindful processes (5). In the inter-professional dialogues, the following principles will underpin the process:

* All partners are experts with various professional experiences,
* Power differentials among partners are acknowledged and sensitively addressed,
* All partners discuss potential benefits and harm of the innovation, research and implementation strategy,
* The process is capacity-building for everyone and encompasses opportunities for mutual learning (4).

DESIGN This is a mixed methods prospective controlled implementation study with an embedded process evaluation. Two similar sized surgical departments will be included; one will be selected as experimental department and the other, as the control. In addition to standard education on HH the experimental ward will participate in an iKT intervention

Participants

1. Leaders and staff at two orthopaedic OR departments within two similar sized university hospitals in the western region of Sweden and Skåne will be invited to take part in the study. Each OR performs approximately 800-900 trauma induced acute hip surgeries annually. One will be selected as the study department and one as the control; approximately 135 persons are employed on each department. Of these, 75% are anaesthetic providers (physicians, nurses and nurse assistants). Both the experimental and the control OR will receive the hospital's standard strategy for infection control: audit and feedback, reminders and computerised education on hand hygiene and the same lecture on Infection Control given by the experts in the area.
2. 1500 patients undergoing fracture surgery of the hip will be invited at each site to take part in a registry study on post-operative complications and satisfaction with the care given.

THE INTERVENTION

Components of the intervention will include:

* Two workshops, consisting of educational sessions covering the state of the art regarding person-centeredness, prevention of infections, leadership, and implementation. The educational component and results of pre-studies will work as frameworks for the dialogues between the front-line leaders and the research group. In dialogues the participants will be given the opportunity to reflect on barriers to and enablers of change; and
* The participants will be supported in creating an action plan aimed at facilitating the anaesthesia providers' change of practice by "1) support, visibility and communication; (2) creating a positive milieu through vision, role modelling and change; and (3) influencing organisational structures and processes through resources, policies and monitoring"(6). The action plan will be executed over 6 months and include 6-8 learning laboratories, led by clinical leaders and facilitated by researchers.

OUTCOME Primary outcome: Process evaluation: Assessing, dose, reach fidelity, acceptability, feasibility and unforeseen consequences of the implementation strategy Secondary outcomes: a) The application of hand hygiene and aseptic techniques during invasive procedures b) Complications after hip surgery

DATA COLLECTION

Process evaluation:

A key element in this project is the process evaluation assessing acceptability, feasibility and unforeseen consequences of the implementation through interviews and ethnographic fieldwork. Ethnographic fieldwork (7) is particularly suited to understanding culture and complexity and finding explanations of why and how specific intervention strategies have failed or succeeded. Participant observations (8) will be made throughout the implementation process. The purpose of using this method is to capture talks and events in relation to the implementation strategies and to understand basic assumptions regarding team-work and patient safety strategies the OR. Attention will be paid to practices that may work as barriers to, and enablers for change. In addition, purposively selected key staff and informal leaders of all professional categories (to ensure maximum variation) will be asked in interviews to give their perspectives on the implementation strategies and activities. The interviews will be audio-taped and transcribed verbatim. In addition to the ethnographic method, structured observations will be used to determine the "dose" of the intervention components given and received, as well as fidelity to the intervention (9).

The use of of hand hygiene/aseptic technique:

The direct observation of hand hygiene is regarded as the gold standard and will be used in this study (10). Adherence to hand hygiene guidelines and aseptic techniques will be measured using a pre-tested and modified version of the World Health Organisation's observational tool (11). The form has been modified to match the OR context (12). An opportunity for hand hygiene is defined as a situation requiring hand disinfection in accordance with national and local guidelines (13). A hand hygiene application is defined as the use of an alcohol-based hand rub in relation to an opportunity. The amount of product used and the duration of its application will not be recorded. Adherence will be recorded in relation to professional category and type of indication. Based on power estimation of 90% power with an alpha level of 5% and an estimated difference before and after the intervention of 10% between the study sites and time periods, 100 care procedures requiring HH and AT will be observed at each time point for each department

Pre-intervention data will be collected in the experimental and the control wards in close connection with the intervention. Post-intervention data will be collected 6 and 12 months after the completed leadership intervention.

Postoperative complications:

The nurses responsible for the discharge will, after on informed consent collect information, from the patients' medical chart on post-operative urinary- and respiratory tract infections, bloodstream and surgical wound infections, pressure-ulcers and confusion. A research assistant will perform chard audits on every 20th included patient to validate data.

Six weeks and 12 months after discharge the patients will be sent by regular mail a survey on patient satisfaction and treatment with antibiotics for wound infection.

Data analysis Interviews and field notes: Inductive content analysis will be used for analysis of qualitative data derived from interviews and participant observations. The texts will be read and re-read to obtain a full understanding and gain a sense of the whole. Meaning units will be extracted, condensed, and labelled with a code, with the aim of the study kept in mind. The code assigned reflected the meaning unit and serves as a tool for viewing the data in a new way. The codes will be compared and grouped into sub-themes. This analysis will continue by interpreting the underlying meaning in relation to time and context with the support of the theoretical framework.

Observational and registry data: The types of statistics used in data analysis will be driven by the level of the data and its distribution. Descriptive statistics will be used to summarize data on AT and inferential statistics used for comparisons between groups and time periods.

Ethics The study will be conducted with approval by the Regional Ethics Review Board in Gothenburg, Sweden. Informed consent will be obtained from the ward managers prior to observation. The project will be conducted in line with the four principal requirements of the Helsinki Declaration; autonomy, non-malfeasance, beneficence, and justice (54). Both oral and written information will be given to the participants and written consent will be sought (appendix 4:1-3). In those cases when potential participating patients suffer from conditions that impede their possibilities to give informed consent, their next of kin will be asked to consider giving consent for participation. All data will be analyzed and reported on group lever. The participant's confidentiality and privacy will be maintained.

ELIGIBILITY:
Inclusion Criteria:

* All staff currently working at the intervention site and control site are eligibly for inclusion

All patient that are undergoing hip fracture surgery at the control and study site and have given informed consent

Exclusion Criteria:

* ongoing infection before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Surgical site infections | 1 year
  At discharge, after 6 weeks and 1 year data will be collect on post-operative infections.

SECONDARY OUTCOMES:
Hand hygiene and Aseptic techniques | At baseline, 6, 12 and 18 month after the start of the intervention
  Adherence to hand hygiene guidelines and aseptic techniques will be measured using a pre-tested and modified version of the World Health Organisation's observational tool (11). The form has been modified to match the OR context (12). An opportunity for hand hygiene is defined as a situation requiring hand disinfection in accordance with national and local guidelines (13). A hand hygiene application is defined as the use of an alcohol-based hand rub in relation to an opportunity. The amount of product used and the duration of its application will not be recorded. Adherence will be recorded in relation to professional category and type of indication. Based on power estimation of 90% power with an alpha level of 5% and an estimated difference before and after the intervention of 10% between the study sites and time periods, 100 care procedures requiring HH and AT will be observed at each time point for each department

OTHER OUTCOMES:
Process evaluation | 1 year
  Process data will be collected using structured observations and ethnographic fieldwork

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska Academy, University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Erichsen Andersson A, Gillespie BM, Karlsson M, Malchau H, Nellgard B, Wikstrom E, Rogmark C, Tillander J. Reduction of early surgical site and other care related infections in 3553 hip fracture patients: lessons learned from the 5-year Safe Hands project. Antimicrob Resist Infect Control. 2022 Sep 5;11(1):113. doi: 10.1186/s13756-022-01153-4. PMID 36064457
- [Derived] Erichsen Andersson A, Frodin M, Dellenborg L, Wallin L, Hok J, Gillespie BM, Wikstrom E. Iterative co-creation for improved hand hygiene and aseptic techniques in the operating room: experiences from the safe hands study. BMC Health Serv Res. 2018 Jan 4;18(1):2. doi: 10.1186/s12913-017-2783-1. PMID 29301519